CLINICAL TRIAL: NCT04829409
Title: The Effects of Ultrasound-guided Mid-point Transverse Process to Pleura Block, Erector Spinae Plane Block and Paravertebral Block on Postoperative Pain in Video-assisted Thoracic Surgery
Brief Title: The Effects of Three Different Ultrasound-guided Nerve Blocks in VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJMZK20210301
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Thoracic Anesthesia; Nerve Block; Pain, Acute
Keywords: ultrasound-guided nerve block; postoperative pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- paravertebral block (Active Comparator): Patients receive ultrasound-guided paravertebral block
  Interventions: Procedure: Paravertebral block
- ESP block (Active Comparator): Patients receive ultrasound-guided erector spinae plane (ESP) block
  Interventions: Procedure: ESP block
- MTP block (Experimental): Patients receive ultrasound-guided mid-point transverse process to pleura (MTP) block
  Interventions: Procedure: MTP block

INTERVENTIONS:
Procedure: Paravertebral block — Patients receive ultrasound-guided paravertebral block
  Arms: paravertebral block
Procedure: ESP block — Patients receive ultrasound-guided erector spinae plane (ESP) block
  Arms: ESP block
Procedure: MTP block — Patients receive ultrasound-guided mid-point transverse process to pleura (MTP) block
  Arms: MTP block

SUMMARY:
Ultrasound-guided mid-point transverse process to pleura block, erector spinae plane block and paravertebral block are three different methods of nerve block, used for relieving postoperative pain in thoracic anesthesia. This study is to compare them on block effects, postoperative pain and analgesic consumption in video-assisted thoracic surgery.

DETAILED DESCRIPTION:
Ultrasound-guided nerve block is an important part of multi-mode analgesia to decrease the consumption of opioids. Thoracic paravertebral block is considered as an ideal regional analgesic choice for video-assisted thoracic surgery, but it still has some side effects, such as pneumothorax, vascular injury, especially for novices. Recent years, ultrasound-guided mid-point transverse process to pleura block and erector spinae plane block are reported for thoracic surgery. The insertion depth in these two methods is more superficial than traditional paravertebral block. They could have less side effects. Therefore, we design a randomised control study to compare them on block effects, postoperative pain and analgesic consumption in video-assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* selective lobetomy under VATS
* ASA classfication 1-3

Exclusion Criteria:

* history of thoracic surgery
* double lateral VATS
* allergy to local anesthetics
* coagulation disorders
* severe heart diseases, hepatic or renal insufficiency
* a history of chronic pain or chronic opioid use
* psychiatric disease or uncooperative
* BMI>28 kg/m2
* VATS transfered to open thoractomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
postoperative morphine consumption | postoperative 24 hours
  The dose is according to the record from PCA pump

SECONDARY OUTCOMES:
Pain score at rest | at 0, 8, 24 hour after surgery
  measured by VAS (0-10)
Pain score while coughing | at 0, 8, 24 hour after surgery
  measured by VAS (0-10)

OTHER OUTCOMES:
block level | 20 minutes after block
  measured by pin-prick at clavicle midline
intraoperative analgesic comsumption | intraoperative, from induction to emergence from anesthesia
  the dose of sufentanil, remifentanil

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, MD,PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China